CLINICAL TRIAL: NCT02201108
Title: A Two Year, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Trial to Evaluate Efficacy, Safety, Tolerability, and Pharmacokinetics of Teriflunomide Administered Orally Once Daily in Pediatric Patients With Relapsing Forms of Multiple Sclerosis Followed by an Open-Label Extension
Brief Title: Efficacy, Safety and Pharmacokinetics of Teriflunomide in Pediatric Patients With Relapsing Forms of Multiple Sclerosis
Acronym: TERIKIDS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC11759; U1111-1124-0983 (Registry Identifier: ICTRP); 2011-005249-12 (EudraCT Number)
Record Dates: First submitted 2014-07-17; First posted 2014-07-25 (Estimated); Results first posted 2020-11-30 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — teriflunomide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (2):
- Placebo (Placebo Comparator): Matching placebo tablets
  Interventions: Drug: Placebo
- Teriflunomide (Experimental): Teriflunomide oral tablet, three dosages (3.5, 7 or 14 mg) to reach 14 mg adult equivalent
  Interventions: Drug: Teriflunomide

INTERVENTIONS:
Drug: Teriflunomide — Pharmaceutical form:film-coated tablet, Route of administration: oral
  Other Names: AUBAGIO, HMR1726
  Arms: Teriflunomide
Drug: Placebo — Pharmaceutical form:tablet, Route of administration: oral
  Arms: Placebo

SUMMARY:
Primary Objective:

To assess the effect of teriflunomide in comparison to placebo on disease activity measured by time to first clinical relapse after randomization in children and adolescents 10 to 17 years of age with relapsing forms of multiple sclerosis (MS).

Secondary Objective:

* To assess the effect of teriflunomide in comparison to placebo on disease activity/progression measured by brain magnetic resonance imaging (MRI) and on cognitive function.
* To evaluate the safety and tolerability of teriflunomide in comparison to placebo.
* To evaluate the pharmacokinetics (PK) of teriflunomide.

DETAILED DESCRIPTION:
The study duration included a screening period up to 4 weeks, a double-blind treatment period of up to 96 weeks, an open-label period which included the remainder of the initial 96 weeks, where applicable, and a 96-week extension, i.e., up to a maximum of 192 weeks after randomization. There was a follow-up period of 4 weeks for participants discontinuing treatment.

Within the 96 weeks double-blind treatment period, the first 4 weeks were PK run-in phase in which PK samples (blood samples) were collected from participants and then 4 weeks of analysis (no samples drawn). The PK run-in phase (total 8 weeks) was intended to provide individual PK parameters to allow the dose adjustment to the 14 milligrams (mg) adult-equivalent dose for the rest of the study.

Participants who experienced a relapse after the PK run-in phase (8 weeks) and confirmed by the Relapse Adjudication Panel and participants who fulfilled MRI criteria (high number of new lesions at weeks 36, 48 or 72 compared to previous images) had the option to continue in an open-label teriflunomide treatment arm up to 192 weeks from randomization.

An optional additional extension period was available for young participants with teriflunomide until the participants are 18 years old and/or able to switch to commercial product, whichever comes first.

ELIGIBILITY:
* Participants with relapsing MS were eligible. Participants who met the criteria of MS based on McDonald criteria 2010 and International Pediatric Multiple Sclerosis Study Group (IPMSSG) criteria for pediatric MS, version of 2012 and had:

  * at least one relapse (or attack) in the 12 months preceding screening or,
  * at least two relapses (or attack) in the 24 months preceding screening.
* Less than 18 years of age and greater than or equal to (>=) 10 years of age at randomization. Specific for the Russian Federation from 18 December 2014 to 26 July 2016, less than or equal to 17 years of age and >= 13 years of age at randomization.
* Signed informed consent/assent obtained from participant and participant's legal representative (parents or guardians) according to local regulations.

Exclusion criteria:

* Expanded disability status scale score greater than 5.5 at screening or randomization visits.
* Relapse within 30 days prior to randomization.
* Treated with:

  * glatiramer acetate, interferons, or dimethyl fumarate within 1 month prior to randomization.
  * fingolimod, or intravenous immunoglobulins within 3 months prior to randomization.
  * natalizumab, other immunosuppressant or immunomodulatory agents such as cyclophosphamide, azathioprine, cyclosporine, methotrexate, mycophenolate, within 6 months prior to randomization.
  * cladribine or mitoxantrone within 2 years prior to randomization.
* Treated with alemtuzumab at any time.
* History of human immunodeficiency virus infection.
* Contraindication for MRI.
* Pregnant or breast-feeding females or those who plan to become pregnant during the study.
* Female participants of child-bearing potential not using highly effective contraceptive method (contraception in both female and male was required).

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 166 (Actual)
Dates: Start 2014-07-16 (Actual); Primary Completion 2019-10-25 (Actual); Study Completion 2024-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (57):
- United States (4):
  - North Central Neurology Associates, PC Site Number : 840003, Cullman, Alabama
  - Axiom Clinical Research of Florida Site Number : 840012, Tampa, Florida
  - Massachusetts General Hospital Site Number : 840002, Boston, Massachusetts
  - Raleigh Neurology Associates Site Number : 840004, Raleigh, North Carolina
- Belgium (2):
  - Investigational Site Number : 056002, Ghent
  - Investigational Site Number : 056001, Leuven
- Investigational Site Number : 100001, Sofia, Bulgaria
- Investigational Site Number : 124001, Calgary, Alberta, Canada
- China (12):
  - Investigational Site Number : 156001, Beijing
  - Investigational Site Number : 156002, Beijing
  - Investigational Site Number : 156010, Beijing
  - Investigational Site Number : 156006, Changchun
  - Investigational Site Number : 156007, Changsha
  - Investigational Site Number : 156008, Chengdu
  - Investigational Site Number : 156005, Chongqing
  - Investigational Site Number : 156012, Guangzhou
  - Investigational Site Number : 156003, Shanghai
  - Investigational Site Number : 156004, Shanghai
  - Investigational Site Number : 156011, Shijiazhuang
  - Investigational Site Number : 156009, Taiyuan
- Investigational Site Number : 233001, Tallinn, Estonia
- France (4):
  - Investigational Site Number : 250001, Le Kremlin-Bicêtre
  - Investigational Site Number : 250002, Lyon
  - Investigational Site Number : 250003, Rennes
  - Investigational Site Number : 250005, Toulouse
- Greece (2):
  - Investigational Site Number : 300002, Athens
  - Investigational Site Number : 300001, Thessaloniki
- Israel (2):
  - Investigational Site Number : 376001, Jerusalem
  - Investigational Site Number : 376003, Tel Litwinsky
- Investigational Site Number : 422001, Beirut, Lebanon
- Investigational Site Number : 440001, Kaunas, Lithuania
- Morocco (2):
  - Investigational Site Number : 504004, Fes
  - Investigational Site Number : 504005, Marrakesh
- Investigational Site Number : 528001, Rotterdam, Netherlands
- North Macedonia (2):
  - Investigational Site Number : 807002, Shtip
  - Investigational Site Number : 807001, Skopje
- Investigational Site Number : 620001, Coimbra, Portugal
- Russia (5):
  - Investigational Site Number : 643001, Moscow
  - Investigational Site Number : 643003, Nizhny Novgorod
  - Investigational Site Number : 643004, Novosibirsk
  - Investigational Site Number : 643005, Saint Petersburg
  - Investigational Site Number : 643002, Saint Petersburg
- Investigational Site Number : 688002, Belgrade, Serbia
- Investigational Site Number : 724002, Murcia, Spain
- Tunisia (3):
  - Investigational Site Number : 788001, Manouba
  - Investigational Site Number : 788002, Sfax
  - Investigational Site Number : 788004, Sfax
- Turkey (Türkiye) (6):
  - Investigational Site Number : 792002, Ankara
  - Investigational Site Number : 792001, Ankara
  - Investigational Site Number : 792006, Istanbul
  - Investigational Site Number : 792003, Istanbul
  - Investigational Site Number : 792008, Izmir
  - Investigational Site Number : 792007, Izmir
- Ukraine (2):
  - Investigational Site Number : 804001, Kharkiv
  - Investigational Site Number : 804002, Kharkiv
- United Kingdom (2):
  - Investigational Site Number : 826001, London, London, City of
  - Investigational Site Number : 826003, Birmingham

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Chitnis T, Banwell B, Kappos L, Arnold DL, Gucuyener K, Deiva K, Saubadu S, Hu W, Benamor M, Le-Halpere A, Truffinet P, Tardieu M. Teriflunomide in pediatric patients with relapsing multiple sclerosis: Open-label extension of TERIKIDS. Mult Scler. 2024 Jun;30(7):833-842. doi: 10.1177/13524585241242050. Epub 2024 Apr 15. PMID 38619037
- [Derived] Kuhle J, Chitnis T, Banwell B, Tardieu M, Arnold DL, Rawlings AM, Geertsen SS, Lublin AL, Saubadu S, Truffinet P, Kappos L. Plasma neurofilament light chain in children with relapsing MS receiving teriflunomide or placebo: A post hoc analysis of the randomized TERIKIDS trial. Mult Scler. 2023 Mar;29(3):385-394. doi: 10.1177/13524585221144742. Epub 2023 Jan 12. PMID 36632983
- [Derived] Chitnis T, Banwell B, Kappos L, Arnold DL, Gucuyener K, Deiva K, Skripchenko N, Cui LY, Saubadu S, Hu W, Benamor M, Le-Halpere A, Truffinet P, Tardieu M; TERIKIDS Investigators. Safety and efficacy of teriflunomide in paediatric multiple sclerosis (TERIKIDS): a multicentre, double-blind, phase 3, randomised, placebo-controlled trial. Lancet Neurol. 2021 Dec;20(12):1001-1011. doi: 10.1016/S1474-4422(21)00364-1. PMID 34800398

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 57 active centers in 21 countries. A total of 185 participants were screened between 16 July 2014 and 27 December 2017, of which 166 participants were enrolled and randomized. A total of 19 participants failed screening mainly due to meeting exclusion criteria.
Pre-assignment Details: Participants were randomly assigned to receive either teriflunomide or placebo in a 2:1 ratio via Interactive Voice Response System. Randomization was stratified by the country and participant's pubertal status.
Groups:
- Placebo/Teriflunomide: Participants received Placebo matching to teriflunomide tablet orally once daily for 96 weeks in double blind (DB) treatment period. After completion of DB period, eligible participants entered in open label (OL) period and received 1 teriflunomide tablet, 3.5 milligrams (mg) (in case of body weight [BW] up to 40 kilograms [kg]) or 7 mg (BW greater than [>] 40 kg) for first 8 weeks. After 8 weeks if individual predicted PK parameter was less than or equal to (<=) 95th percentile of adult range after 7 mg once daily, then participants received 1 tablet of 7 mg teriflunomide daily (for BW up to 40 kg) or 1 tablet of 14 mg teriflunomide daily (for BW>40 kg) in the OL period for additional 96 weeks (i.e., up to Week 192). If individual predicted PK parameters >95th percentile of adult range then participant received 1 tablet of 3.5 mg teriflunomide daily (for BW up to 40 kg) or 1 tablet of 7 mg teriflunomide daily (for BW >40 kg).The adult range (5th-95th percentile) of predicted steady state PK parameters for a 7 mg dose was defined as maximum concentration observed (Cmax) ranging from 8.03 to 49.10 micrograms per milliliter (mcg/mL) and area under the curve from time 0 hour to 24 hours (AUC0-24) ranging from 184 to 1160 micrograms*hour per milliliter (mcg*h/mL).
- Teriflunomide/Teriflunomide: Participants received 1 teriflunomide tablet, 3.5 mg (in case of BW up to 40 kg) or 7 mg (in case of BW >40 kg) orally once daily for 8 weeks. After 8 weeks, based on individual predicted PK parameters, teriflunomide was administered in following manner up to 96 weeks: if predicted PK parameters <= 95th percentile of adult range after 7 mg once daily, then participants received 1 tablet of 7 mg teriflunomide daily (for BW up to 40 kg) or 1 tablet of 14 mg teriflunomide daily (for BW >40 kg); or if individual predicted PK parameters >95th percentile of adult range then participants received 1 tablet of 3.5 mg teriflunomide daily (for BW up to 40 kg) or 1 tablet of 7 mg teriflunomide daily (for BW >40 kg). The adult range (5th - 95th percentile) of predicted steady state PK parameters for a 7 mg dose was defined as Cmax ranging from 8.03 to 49.10 mcg/mL and AUC0-24 ranging from 184 to 1160 mcg*h/mL. After completion of DB period, eligible participants entered in OL period and continued receiving teriflunomide at the same dose in the OL period for additional 96 weeks (i.e., up to Week 192).
- Teriflunomide: Participants who were not adults when they completed the 192-week OL period were offered an optional additional extension period to receive 1 teriflunomide tablet 14 mg daily (or every other day if BW was <40 kg) until they became adults or until they were able to switch to the commercial product, whichever came first.
Period: Double-blind Period (up to Week 96)
Arm/Group | Placebo/Teriflunomide | Teriflunomide/Teriflunomide | Teriflunomide
Started (Randomized and treated participants.) | 57 | 109 | 0
Completed | 53 | 102 | 0
Not Completed | 4 | 7 | 0
Not completed — Adverse Event | 0 | 6 | 0
Not completed — Lack of Efficacy | 2 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0
Period: Open Label Period (up to Week 192)
Arm/Group | Placebo/Teriflunomide | Teriflunomide/Teriflunomide | Teriflunomide
Started (Post completion of DB treatment period, only eligible participants entered OL treatment period.) | 52 | 100 | 0
Completed | 31 | 73 | 0
Not Completed | 21 | 27 | 0
Not completed — Lack of Efficacy | 10 | 14 | 0
Not completed — Poor compliance to protocol | 0 | 1 | 0
Not completed — Other reason | 4 | 7 | 0
Not completed — Adverse Event | 7 | 5 | 0
Period: Extension Period (Up to Week 492)
Arm/Group | Placebo/Teriflunomide | Teriflunomide/Teriflunomide | Teriflunomide
Started (Post completion of OL treatment period, only eligible participants entered extension period.) | 0 | 0 | 27
Completed | 0 | 0 | 24
Not Completed | 0 | 0 | 3
Not completed — Adverse Event | 0 | 0 | 2
Not completed — Poor compliance to protocol | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all randomized participants.
Groups:
- Placebo/Teriflunomide: Participants received Placebo matching to teriflunomide tablet orally once daily for 96 weeks in DB treatment period. After completion of DB period, eligible participants entered in OL period and received 1 teriflunomide tablet, 3.5 mg (in case of BW up to 40 kg) or 7 mg (in case of BW >40 kg) for first 8 weeks. After 8 weeks if individual predicted PK parameter was <= 95th percentile of adult range after 7 mg once daily, then participants received 1 tablet of 7 mg teriflunomide daily (for BW up to 40 kg) or 1 tablet of 14 mg teriflunomide daily (for BW>40 kg) in the OL period for additional 96 weeks (i.e., up to Week 192). If individual predicted PK parameters >95th percentile of adult range then participant received 1 tablet of 3.5 mg teriflunomide daily (for BW up to 40 kg) or 1 tablet of 7 mg teriflunomide daily (for BW >40 kg). The adult range (5th-95th percentile) of predicted steady state PK parameters for a 7 mg dose was defined as Cmax ranging from 8.03 to 49.10 mcg/mL and AUC0-24 ranging from 184 to 1160 mcg*h/mL.
- Total: Total of all reporting groups
Arm/Group | Placebo/Teriflunomide | Teriflunomide/Teriflunomide | Total
Number analyzed (Participants) | 57 | 109 | 166
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.7 (2.1) | 14.6 (2.0) | 14.6 (2.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 72 | 111
  Male | 18 | 37 | 55
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Caucasian/White | 42 | 75 | 117
  Race: Black | 1 | 4 | 5
  Race: Asian/Oriental | 12 | 25 | 37
  Race: Other | 2 | 5 | 7

OUTCOME MEASURES:

1. Primary Outcome: Time to First Confirmed Clinical Relapse
Description: Time to first clinical relapse was defined as the duration (in weeks) between randomization and first confirmed clinical relapse. Clinical relapses were defined as new or recurrent neurological symptoms not associated with fever or infection, lasting at least 24 hours, and accompanied by new objective neurological findings upon neurological examination and documented by a standardized, quantified functional system score (FSSs) which included 8 items and items were rated on different scales: brain stem, cerebellar and cerebral functions rated on a scale of 0 to 5; visual, pyramidal, sensory and bowel/bladder rated on a scale of 0 to 6 and ambulation on a scale of 0 to 12, where higher score in each scale indicated worsened neurological function. Confirmed clinical relapse were reviewed and confirmed by an independent Relapse Adjudication Panel (RAP). A participant without confirmed clinical relapse, was considered as clinical relapse free until the end of Week 96.
Time Frame: Baseline up to Week 96
Population: Analysis was performed on Intent-to-treat (ITT) population, which consisted of all randomized participants analyzed according to the treatment allocated by randomization.
Measure: Median (Full Range); unit: weeks
Groups:
- Double-Blind Treatment Period: Placebo: Participants received Placebo matching to teriflunomide tablet orally once daily for 96 weeks in DB period.
- Double-Blind Treatment Period: Teriflunomide: Participants received 1 teriflunomide tablet, 3.5 mg (in case of BW up to 40 kg) or 7 mg (in case of BW >40 kg) orally once daily for 8 weeks. After 8 weeks, based on individual predicted PK parameters, teriflunomide was administered in following manner up to 96 weeks: if predicted PK parameters <= 95th percentile of adult range after 7 mg once daily: 1 tablet of 7 mg teriflunomide daily (for BW up to 40 kg) or 1 tablet of 14 mg teriflunomide daily (for BW >40 kg); or if individual predicted PK parameters >95th percentile of adult range then participants received 1 tablet of 3.5 mg teriflunomide daily (for BW up to 40 kg) or 1 tablet of 7 mg teriflunomide daily (for BW >40 kg). The adult range (5th - 95th percentile) of predicted steady state PK parameters for a 7 mg dose was defined as Cmax ranging from 8.03 to 49.10 mcg/mL and AUC0-24 ranging from 184 to 1160 mcg*h/mL in DB period.
Arm/Group | Double-Blind Treatment Period: Placebo | Double-Blind Treatment Period: Teriflunomide
Number analyzed (Participants) | 57 | 109
weeks | 39.14 [0.1 to 98.0] | 75.29 [0.1 to 98.7]
Statistical Analysis 1: Comparison: Double-Blind Treatment Period: Placebo vs Double-Blind Treatment Period: Teriflunomide; Test type: Superiority; p = 0.2949, Stratified Log-Rank test — Threshold for significance was < 0.05; P-value derived from log-rank test with stratification of region and pubertal status; Hazard Ratio (HR) = 0.657, 95% CI 2-sided [0.388 to 1.113] — Hazard ratio was estimated using a Cox proportional-hazards model with factors for treatment group, region, pubertal status, age, and number of relapses in the year prior to randomization as covariates and with robust variance estimation

2. Secondary Outcome: Probability of Participants Who Were Clinical Relapse Free at Weeks 24, 48, 72, 96, 120, 144, 168 and 192
Description: Participant was considered free of clinical relapse if the participant had no confirmed clinical relapse before treatment discontinuation/completion in 192 weeks treatment period. Clinical relapses: new/recurrent neurological symptoms not associated with fever/infection, lasted at least 24 hours, and accompanied by new objective neurological findings upon neurological examination and documented by standardized, quantified FSSs which included 8 items: rated on different scales: brain stem, cerebellar and cerebral functions rated on scale of 0 to 5; visual, pyramidal, sensory and bowel/bladder rated on scale of 0 to 6 & ambulation on scale of 0 to 12, where higher score in each scale indicated worsened neurological function. New/recurrent symptoms occurred less than 30 days following onset of relapse were considered part of same relapse. Probability of participants who were clinical relapse free at specified weeks were estimated by Kaplan-Meier method and reported.
Time Frame: Weeks 24, 48, 72, 96, 120, 144, 168 and 192
Population: Analysis was performed on efficacy population which included all participants enrolled and treated with at least 1 dose of teriflunomide in OL period analyzed according to the treatment group allocated by randomization in the DB period.
Measure: Number (95% Confidence Interval); unit: probability of relapse free participants
Groups:
- Teriflunomide/ Teriflunomide: Participants received 1 teriflunomide tablet, 3.5 mg (in case of BW up to 40 kg) or 7 mg (in case of BW >40 kg) orally once daily for 8 weeks. After 8 weeks, based on individual predicted PK parameters, teriflunomide was administered in following manner up to 96 weeks: if predicted PK parameters <= 95th percentile of adult range after 7 mg once daily, then participants received 1 tablet of 7 mg teriflunomide daily (for BW up to 40 kg) or 1 tablet of 14 mg teriflunomide daily (for BW >40 kg); or if individual predicted PK parameters >95th percentile of adult range then participants received 1 tablet of 3.5 mg teriflunomide daily (for BW up to 40 kg) or 1 tablet of 7 mg teriflunomide daily (for BW >40 kg). The adult range (5th - 95th percentile) of predicted steady state PK parameters for a 7 mg dose was defined as Cmax ranging from 8.03 to 49.10 mcg/mL and AUC0-24 ranging from 184 to 1160 mcg*h/mL. After completion of DB period, eligible participants entered in OL period and continued receiving teriflunomide at the same dose in the OL period for additional 96 weeks (i.e., up to Week 192).
Arm/Group | Placebo/Teriflunomide | Teriflunomide/ Teriflunomide
Number analyzed (Participants) | 52 | 100
probability of relapse free participants
  Week 24 | 0.750 [0.609 to 0.846] | 0.820 [0.730 to 0.883]
  Week 48 | 0.596 [0.451 to 0.715] | 0.700 [0.600 to 0.780]
  Week 72 | 0.519 [0.377 to 0.644] | 0.630 [0.528 to 0.716]
  Week 96 | 0.442 [0.305 to 0.571] | 0.600 [0.497 to 0.688]
  Week 120 | 0.404 [0.271 to 0.533] | 0.570 [0.467 to 0.660]
  Week 144 | 0.365 [0.238 to 0.494] | 0.540 [0.437 to 0.631]
  Week 168 | 0.365 [0.238 to 0.494] | 0.518 [0.416 to 0.611]
  Week 192 | 0.365 [0.238 to 0.494] | 0.518 [0.416 to 0.611]

3. Secondary Outcome: Brain Magnetic Resonance Imaging (MRI) Assessment: Number of New or Enlarged T2 Lesions Per MRI Scan
Description: Number of new or enlarged T2 lesions per scan was defined as the total number of new or enlarged T2 lesion that occurred during the 192 weeks treatment period divided by the total number of scans performed during 192 weeks. To account for the different numbers of scans performed among the participants, a negative binomial regression model with robust variance estimation was used. The model included the total number of new or enlarged T2-lesions as the response variable, with treatment group, region, pubertal status and age as covariates and log-transformed number of scans as an offset variable.
Time Frame: Baseline up to Week 192
Population: Analysis was performed on efficacy population.
Measure: Number (95% Confidence Interval); unit: lesions per scan
Arm/Group | Placebo/Teriflunomide | Teriflunomide/ Teriflunomide
Number analyzed (Participants) | 52 | 100
lesions per scan | 11.087 [6.586 to 18.662] | 5.664 [3.417 to 9.389]
Statistical Analysis 1: Comparison: Placebo/Teriflunomide vs Teriflunomide/ Teriflunomide; Test type: Other; Relative risk ratio = 0.511, 95% CI 2-sided [0.343 to 0.762]

4. Secondary Outcome: Brain Magnetic Resonance Imaging Assessment: Number of T1 Gadolinium (Gd)-Enhancing T1 Lesions Per MRI Scan
Description: The number of T1 Gd-Enhancing lesions per scan was defined as the total number of Gd-enhancing lesions that occurred during the 192 weeks treatment period divided by the total number of scans performed during 192 weeks. To account for the different number of scans performed among the participants, a negative binomial regression model with robust variance estimation was used. The model included the total number of T1-lesions as the response variable, with treatment group, region, pubertal status and age as covariates and log-transformed number of scans as an offset variable.
Time Frame: Baseline up to Week 192
Population: Analysis was performed on efficacy population.
Measure: Number (95% Confidence Interval); unit: lesions per scan
Arm/Group | Placebo/Teriflunomide | Teriflunomide/ Teriflunomide
Number analyzed (Participants) | 52 | 100
lesions per scan | 2.686 [1.263 to 5.712] | 1.532 [0.624 to 3.762]
Statistical Analysis 1: Comparison: Placebo/Teriflunomide vs Teriflunomide/ Teriflunomide; Test type: Other; Relative risk ratio = 0.57, 95% CI 2-sided [0.331 to 0.983]

5. Secondary Outcome: Brain Magnetic Resonance Imaging Assessment: Change From Baseline in Volume of T2 Lesions at Weeks 24, 36, 48, 72, 96, 144 and 192
Description: Volume of T2 lesions was measured by MRI scan.
Time Frame: Baseline, DB period: Weeks 24, 36, 48, 72 and 96; OL period: Weeks 48, 96, 144 and 192
Population: Analysis was performed on efficacy population. Here, 'overall number of participants analyzed' = participants evaluable for this outcome measure and 'number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Placebo/Teriflunomide | Teriflunomide/ Teriflunomide
Number analyzed (Participants) | 52 | 98
milliliters
  DB Period: Week 24: number analyzed (Participants) | 40 | 88
  DB Period: Week 24 | 3.0 (7.0) | 0.5 (1.8)
  DB Period: Week 36: number analyzed (Participants) | 19 | 39
  DB Period: Week 36 | 4.6 (11.7) | 4.4 (21.3)
  DB Period: Week 48: number analyzed (Participants) | 21 | 68
  DB Period: Week 48 | 0.5 (0.6) | -0.2 (3.4)
  DB Period: Week 72: number analyzed (Participants) | 16 | 59
  DB Period: Week 72 | 1.2 (1.6) | 0.1 (1.9)
  DB Period: Week 96: number analyzed (Participants) | 14 | 51
  DB Period: Week 96 | 0.9 (1.4) | 0.2 (1.9)
  OL Period: Week 48: number analyzed (Participants) | 51 | 88
  OL Period: Week 48 | 3.0 (9.7) | 0.6 (8.8)
  OL Period: Week 96: number analyzed (Participants) | 37 | 74
  OL Period: Week 96 | 2.7 (8.1) | 1.9 (4.0)
  OL Period: Week 144: number analyzed (Participants) | 20 | 23
  OL Period: Week 144 | 4.7 (10.7) | 0.4 (17.1)
  OL Period: Week 192: number analyzed (Participants) | 5 | 8
  OL Period: Week 192 | 0.4 (9.4) | -3.6 (30.6)

6. Secondary Outcome: Brain Magnetic Resonance Imaging Assessment: Change From Baseline in Volume of T1 Hypointense Lesions
Description: Volume of T1 hypointense lesions was measured by MRI scan.
Time Frame: Baseline, DB period: Weeks 24, 36, 48, 72 and 96; OL period: Weeks 48, 96, 144 and 192
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Placebo/Teriflunomide | Teriflunomide/ Teriflunomide
Number analyzed (Participants) | 52 | 98
milliliters
  DB Period: Week 24: number analyzed (Participants) | 40 | 88
  DB Period: Week 24 | 0.3 (1.3) | 0.0 (0.7)
  DB Period: Week 36: number analyzed (Participants) | 19 | 39
  DB Period: Week 36 | 0.8 (1.8) | 0.2 (0.8)
  DB Period: Week 48: number analyzed (Participants) | 20 | 68
  DB Period: Week 48 | 0.2 (0.4) | 0.4 (2.9)
  DB Period: Week 72: number analyzed (Participants) | 16 | 58
  DB Period: Week 72 | 0.1 (0.7) | 0.1 (0.6)
  DB Period: Week 96: number analyzed (Participants) | 14 | 50
  DB Period: Week 96 | 0.1 (0.6) | 0.1 (0.7)
  OL Period: Week 48: number analyzed (Participants) | 51 | 86
  OL Period: Week 48 | 0.7 (1.9) | 0.5 (1.4)
  OL Period: Week 96: number analyzed (Participants) | 37 | 73
  OL Period: Week 96 | 1.0 (2.0) | 0.6 (1.9)
  OL Period: Week 144: number analyzed (Participants) | 20 | 22
  OL Period: Week 144 | 2.0 (3.0) | 1.9 (3.4)
  OL Period: Week 192: number analyzed (Participants) | 5 | 8
  OL Period: Week 192 | 4.0 (5.8) | 2.5 (5.7)

7. Secondary Outcome: Brain Magnetic Resonance Imaging Assessment: Number of New T1 Hypointense Lesions Per MRI Scan
Description: The number of new T1 hypointense lesions were obtained from MRI scans.
Time Frame: Baseline up to Week 192
Population: Analysis was performed on efficacy population.
Measure: Number; unit: lesions
Arm/Group | Placebo/Teriflunomide | Teriflunomide/ Teriflunomide
Number analyzed (Participants) | 52 | 100
lesions | 1561 | 1910
Statistical Analysis 1: Comparison: Placebo/Teriflunomide vs Teriflunomide/ Teriflunomide; Test type: Other; Relative risk ratio = 0.498, 95% CI 2-sided [0.296 to 0.836]

8. Secondary Outcome: Brain Magnetic Resonance Imaging Assessment: Percentage of Participants Free of New or Enlarged MRI T2-Lesions
Description: Percentage of participants who were free of new or enlarged T2 lesions at Weeks 24, 48, 72, 96, 144 and 192 were reported.
Time Frame: Baseline, Weeks 24, 48, 72, 96, 144 and 192
Population: Analysis was performed on efficacy population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo/Teriflunomide | Teriflunomide/ Teriflunomide
Number analyzed (Participants) | 52 | 100
percentage of participants
  Week 24 | 86.5 | 86.0
  Week 48 | 32.7 | 25.0
  Week 72 | 15.4 | 17.0
  Week 96 | 15.4 | 16.0
  Week 144 | 11.5 | 14.0
  Week 192 | 7.7 | 9.0

9. Secondary Outcome: Brain Magnetic Resonance Imaging Assessment: Percent Change From Baseline in Brain Volume at Weeks 24, 36, 48, 72, 96, 144 and 192
Description: Percent change from baseline in brain volume (assessed using MRI scans of the Brain) at Weeks 24, 36, 48,72, 96, 144 and 192 was reported.
Time Frame: Baseline, DB period: Weeks 24, 36, 48, 72 and 96; OL period: Weeks 48, 96, 144 and 192
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo/Teriflunomide | Teriflunomide/ Teriflunomide
Number analyzed (Participants) | 52 | 97
percent change
  DB Period: Week 24: number analyzed (Participants) | 38 | 83
  DB Period: Week 24 | -0.3 (0.7) | -0.2 (0.7)
  DB Period: Week 36: number analyzed (Participants) | 17 | 39
  DB Period: Week 36 | -0.7 (0.7) | -0.4 (1.0)
  DB Period: Week 48: number analyzed (Participants) | 20 | 64
  DB Period: Week 48 | -0.6 (1.1) | -0.5 (0.9)
  DB Period: Week 72: number analyzed (Participants) | 16 | 53
  DB Period: Week 72 | -0.9 (1.3) | -0.6 (1.1)
  DB Period: Week 96: number analyzed (Participants) | 13 | 47
  DB Period: Week 96 | -0.9 (1.3) | -0.8 (1.1)
  OL Period: Week 48: number analyzed (Participants) | 43 | 73
  OL Period: Week 48 | -1.4 (1.6) | -1.1 (1.3)
  OL Period: Week 96: number analyzed (Participants) | 33 | 60
  OL Period: Week 96 | -1.8 (1.9) | -1.4 (1.6)
  OL Period: Week 144: number analyzed (Participants) | 16 | 17
  OL Period: Week 144 | -3.1 (2.8) | -2.0 (1.7)
  OL Period: Week 192: number analyzed (Participants) | 4 | 6
  OL Period: Week 192 | -2.2 (1.2) | -3.0 (1.9)

10. Secondary Outcome: Cognitive Assessment: Change From Baseline in Total Number of Correct Substitutions Measured by Symbol Digit Modalities Test (SDMT) at Weeks 24, 48, 72, 96, 120, 144, 168 and 192
Description: SDMT measures the time to pair abstract symbols with specific numbers. It is a simple substitution task that gives the examinee 90 seconds to pair specific numbers with given geometric figures as a measure for screening cognitive impairment. The SDMT score is the number of correct substitution and ranged from 0 (worst outcome) to 110 (best outcome), where higher score indicated better cognitive function.
Time Frame: Baseline, DB period: Weeks 24, 48, 72 and 96; OL period: Weeks 24, 48, 72, 96, 120, 144, 168 and 192
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo/Teriflunomide | Teriflunomide/ Teriflunomide
Number analyzed (Participants) | 51 | 96
score on a scale
  DB Period: Week 24: number analyzed (Participants) | 40 | 85
  DB Period: Week 24 | 5.1 (12.0) | 4.6 (9.1)
  DB Period: Week 48: number analyzed (Participants) | 20 | 64
  DB Period: Week 48 | 7.3 (14.1) | 5.7 (10.3)
  DB Period: Week 72: number analyzed (Participants) | 17 | 58
  DB Period: Week 72 | 6.4 (12.9) | 5.6 (11.5)
  DB Period: Week 96: number analyzed (Participants) | 14 | 52
  DB Period: Week 96 | 8.8 (10.7) | 8.1 (11.1)
  OL Period: Week 24: number analyzed (Participants) | 51 | 91
  OL Period: Week 24 | 6.3 (13.9) | 8.3 (12.3)
  OL Period: Week 48: number analyzed (Participants) | 44 | 88
  OL Period: Week 48 | 6.7 (13.3) | 7.6 (13.0)
  OL Period: Week 72: number analyzed (Participants) | 41 | 76
  OL Period: Week 72 | 8.0 (15.5) | 9.2 (13.0)
  OL Period: Week 96: number analyzed (Participants) | 36 | 73
  OL Period: Week 96 | 7.6 (16.7) | 8.0 (14.8)
  OL Period: Week 120: number analyzed (Participants) | 22 | 28
  OL Period: Week 120 | 3.7 (15.9) | 7.2 (10.3)
  OL Period: Week 144: number analyzed (Participants) | 18 | 19
  OL Period: Week 144 | 6.6 (14.4) | 5.2 (13.0)
  OL Period: Week 168: number analyzed (Participants) | 13 | 15
  OL Period: Week 168 | 3.5 (17.9) | 1.7 (14.0)
  OL Period: Week 192: number analyzed (Participants) | 1 | 4
  OL Period: Week 192 | 12.0 | -0.3 (18.2)

11. Secondary Outcome: Cognitive Assessment: Change From Baseline in Number of Completed Items Measured by Symbol Digit Modalities Test at Weeks 24, 48, 72, 96, 120, 144, 168 and 192
Description: SDMT measures the time to pair abstract symbols with specific numbers. It is a simple substitution task that gives the examinee 90 seconds to pair specific numbers with given geometric figures as a measure for screening cognitive impairment. The SDMT score is the number of completed items and ranged from 0 (worst outcome) to 110 (best outcome), where higher score indicated better cognitive function.
Time Frame: Baseline, DB period: Weeks 24, 48, 72 and 96; OL period: Weeks 24, 48, 72, 96, 120, 144, 168 and 192
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo/Teriflunomide | Teriflunomide/ Teriflunomide
Number analyzed (Participants) | 51 | 96
score on a scale
  DB Period: Week 24: number analyzed (Participants) | 40 | 85
  DB Period: Week 24 | 3.8 (11.7) | 3.6 (9.0)
  DB Period: Week 48: number analyzed (Participants) | 20 | 64
  DB Period: Week 48 | 6.3 (13.8) | 4.7 (10.3)
  DB Period: Week 72: number analyzed (Participants) | 17 | 58
  DB Period: Week 72 | 5.1 (13.4) | 4.5 (11.4)
  DB Period: Week 96: number analyzed (Participants) | 14 | 52
  DB Period: Week 96 | 7.1 (11.2) | 6.9 (11.1)
  OL Period: Week 24: number analyzed (Participants) | 51 | 91
  OL Period: Week 24 | 4.8 (13.5) | 7.1 (12.4)
  OL Period: Week 48: number analyzed (Participants) | 44 | 88
  OL Period: Week 48 | 5.5 (12.8) | 6.4 (13.0)
  OL Period: Week 72: number analyzed (Participants) | 41 | 76
  OL Period: Week 72 | 6.4 (15.4) | 8.1 (12.8)
  OL Period: Week 96: number analyzed (Participants) | 36 | 73
  OL Period: Week 96 | 6.3 (16.6) | 7.6 (12.5)
  OL Period: Week 120: number analyzed (Participants) | 22 | 28
  OL Period: Week 120 | 3.7 (14.7) | 6.3 (11.5)
  OL Period: Week 144: number analyzed (Participants) | 18 | 19
  OL Period: Week 144 | 4.8 (15.1) | 3.7 (13.4)
  OL Period: Week 168: number analyzed (Participants) | 13 | 15
  OL Period: Week 168 | 2.7 (15.5) | -0.3 (15.6)
  OL Period: Week 192: number analyzed (Participants) | 1 | 4
  OL Period: Week 192 | 12.0 | -1.5 (18.3)

12. Secondary Outcome: Cognitive Assessment: Change From Baseline in Brief Visuospatial Memory Test-Revised (BVMT-R) Scores at Weeks 96 and 192
Description: The BVMT consists of three trials in which participants must recall shapes by drawing figures on a blank page (response booklet) after being given the opportunity to memorize the figures (given in BMVT-R form) for 10 seconds. BMVT-R form consists of six figures. Points are awarded based on the accuracy of the drawn figure and by correct placement on the blank page. A minimum of 0 to 12 points/scores are awarded per trial, so a participant can score between 0 and 36 points for all three trials (by adding the points/score from each trial), where higher score indicates better outcome.
Time Frame: Baseline, Weeks 96 and 192
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo/Teriflunomide | Teriflunomide/ Teriflunomide
Number analyzed (Participants) | 31 | 69
score on a scale
  Baseline | 23.8 (7.2) | 24.8 (6.4)
  Change at Week 96: number analyzed (Participants) | 5 | 35
  Change at Week 96 | -0.8 (9.3) | 1.6 (5.3)
  Change at Week 192: number analyzed (Participants) | 16 | 45
  Change at Week 192 | 1.0 (6.9) | 1.2 (5.4)

13. Secondary Outcome: Cognitive Assessment: Change From Baseline in Trail Making Test- Part A (TMT-A) Test Scores (in Seconds) at Week 96 and 192
Description: 'Trail Making Test Part A' is a neuropsychological test of visual attention and task switching. The task requires a participant to 'connect-the-dots' of 25 consecutive numbers (1,2, 3, etc.) in sequential order on a sheet of paper or computer screen. The goal of the participant is to finish the test as quickly as possible, and the time taken to complete the test used as the primary performance metric (in seconds). This is a timed test and the number of seconds to complete the task is recorded. Maximum time allowed is 300 seconds. A lower score indicated better cognitive function.
Time Frame: Baseline, Weeks 96 and 192
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Placebo/Teriflunomide | Teriflunomide/ Teriflunomide
Number analyzed (Participants) | 14 | 29
seconds
  Baseline | 43.4 (24.2) | 47.1 (23.7)
  Change at Week 96: number analyzed (Participants) | 3 | 13
  Change at Week 96 | 8.4 (9.0) | -3.1 (19.5)
  Change at Week 192: number analyzed (Participants) | 8 | 21
  Change at Week 192 | 6.3 (20.7) | -6.6 (17.4)

14. Secondary Outcome: Cognitive Assessment: Change From Baseline in Trail Making Test B (TMT-B) Test Scores (in Seconds) at Weeks 96 and 192
Description: TMT-B is a cognitive test that gives a measure of various aspects of cognitive performance. It is used to measure cognitive fatigue. The test consisted of 25 circles containing 13 sequential numbers (1 to 13) and 12 sequential letters (A to L) positioned. The test evaluates the time (in seconds) to correctly order letters and numbers in alternate order (1, A, 2, B etc.). Maximum time allowed is 300 seconds, where less time/lower score indicated better cognitive function/performance.
Time Frame: Baseline, Weeks 96 and 192
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Placebo/Teriflunomide | Teriflunomide/ Teriflunomide
Number analyzed (Participants) | 14 | 28
seconds
  Baseline | 113.8 (81.5) | 115.0 (44.6)
  Change at Week 96: number analyzed (Participants) | 3 | 13
  Change at Week 96 | -19.8 (33.7) | -29.5 (56.6)
  Change at Week 192: number analyzed (Participants) | 8 | 21
  Change at Week 192 | -37.0 (83.3) | -18.8 (37.3)

15. Secondary Outcome: Cognitive Assessment: Change From Baseline in Beery Visual-motor Integration (BVMI) Scores at Weeks 96 and 192
Description: The Beery VMI is a non-verbal assessment that assessed the extent to which individuals can integrate their visual and motor abilities. The participants were provided with geometric designs ranging from simple line drawings to more complex figures and were asked to copy the designs. The test consisted of 24 figures. One point was scored for each successful copy of drawings and no scoring was given when the participant failed to copy the drawings properly. Each successful copying of drawings was summed up and the total was scored on a scale ranged from 0 to 24, where higher score indicated better visual construction skills/better visual and motor abilities and lower score indicated poor visual construction skills/poor visual and motor abilities.
Time Frame: Baseline, Weeks 96 and 192
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo/Teriflunomide | Teriflunomide/ Teriflunomide
Number analyzed (Participants) | 39 | 82
score on a scale
  Baseline | 26.1 (5.2) | 25.9 (4.0)
  Change at Week 96: number analyzed (Participants) | 10 | 47
  Change at Week 96 | 0.6 (2.4) | -0.4 (4.8)
  Change at Week 192: number analyzed (Participants) | 26 | 58
  Change at Week 192 | 0.1 (5.4) | 0.4 (2.9)

16. Secondary Outcome: Cognitive Assessment: Change From Baseline in Wechsler Abbreviated Scale of Intelligence-II (WASI-II) Vocabulary Total Raw Scores at Weeks 96 and 192
Description: The WASI-II: Vocabulary test is a quick estimate of an individual's level of intellectual functioning which comprised of 31 total items that required the participant to orally define 3 images and 28 words presented both orally and visually. Items 1 to 3 rated on a score of 0 or 1, items 4 and 5 rated on a score of 0 or 2, items 6 to 31 rated on a scale of 0 to 2. Each item score was summed up to derive the total score which ranged from 0 (minimum score) to 59 (maximum score), where higher score indicated better level of intellectual functioning/higher level of intelligence.
Time Frame: Baseline, Weeks 96 and 192
Population: Analysis was performed on efficacy population. Here, "overall number of participants analyzed" = participants evaluable for this outcome measure and 'number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo/Teriflunomide | Teriflunomide/ Teriflunomide
Number analyzed (Participants) | 1 | 3
score on a scale
  Baseline | 39.0 | 34.3 (7.0)
  Change at Week 96: number analyzed (Participants) | 1 | 1
  Change at Week 96 | 5.0 | 4.0
  Change at Week 192: number analyzed (Participants) | 1 | 1
  Change at Week 192 | 3.0 | 5.0

17. Secondary Outcome: Cognitive Assessment: Change From Baseline in Delis-Kaplan Executive Function System (D-KEFS) Letter Fluency Total Correct Raw Score at Weeks 96 and 192
Description: Letter Fluency is a condition measured in the D-KEFS. Participants were asked to name as many words as they can, starting with a specified letter for 60 seconds. The words cannot be names, places, numbers or grammatical variants of previous answers. Repeated answers were not scored as a correct response. There were 3 trials, with 3 different letters. The total number of correct responses was totaled for all 3 trials and a letter fluency score was given. A higher score was considered better. There was no set range as the score depends on how many correct words the participant relays in the given time period.
Time Frame: Baseline, Weeks 96 and 192
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo/Teriflunomide | Teriflunomide/ Teriflunomide
Number analyzed (Participants) | 2 | 6
score on a scale
  Baseline | 32.5 (3.5) | 21.0 (6.0)
  Change at Week 96: number analyzed (Participants) | 1 | 2
  Change at Week 96 | -3.0 | 4.0 (9.9)
  Change at Week 192: number analyzed (Participants) | 1 | 2
  Change at Week 192 | 5.0 | -6.5 (16.3)

18. Secondary Outcome: Cognitive Assessment: Change From Baseline in Delis-Kaplan Executive Function System Category Fluency Total Correct Raw Score at Weeks 96 and 192
Description: Category Fluency is a condition measured in the D-KEFS. It measured participant's ability to generate words from three different categories (e.g., fruits, vegetables and animals), within a minute for each category. Total score was number of correct words for each category with no points for repetitions or non-words. Score ranged from 0 to unlimited, where 0 = low score, higher score indicated better performance.
Time Frame: Baseline, Weeks 96 and 192
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo/Teriflunomide | Teriflunomide/ Teriflunomide
Number analyzed (Participants) | 2 | 6
score on a scale
  Baseline | 28.0 (1.4) | 27.5 (9.2)
  Change at Week 96: number analyzed (Participants) | 1 | 2
  Change at Week 96 | 6.0 | 5.0 (5.7)
  Change at Week 192: number analyzed (Participants) | 1 | 2
  Change at Week 192 | -2.0 | -13.5 (17.7)

19. Secondary Outcome: Cognitive Assessment - Selective Reminding Test (SRT): Change From Baseline in Total Number of Words on Delayed Recall at Weeks 96 and 192
Description: SRT is a test to assess verbal learning and memory. During the administration of the SRT only the examiner and the participant should be in the testing room. A list of twelve words was read aloud by the examiner at a rate of one word per two seconds. The participant is asked to recall all twelve words after a 30 minute delay. Only the words that were missed on the preceding trial were given in the consecutive trial. The total score represented a sum score of total 6 trials, therefore the score range was from 0 to 72. The lower the score the worse the outcome, higher score indicated better recall.
Time Frame: Baseline, Weeks 96 and 192
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo/Teriflunomide | Teriflunomide/ Teriflunomide
Number analyzed (Participants) | 2 | 4
score on a scale
  Baseline | 3.5 (4.9) | 10.0 (1.4)
  Change at Week 96: number analyzed (Participants) | 1 | 2
  Change at Week 96 | 1.0 | -0.5 (2.1)
  Change at Week 192: number analyzed (Participants) | 1 | 1
  Change at Week 192 | 0.0 | 0.0

20. Secondary Outcome: DB: Pharmacokinetics: Steady-state Trough Concentration (Ctrough) of Teriflunomide
Description: Ctrough was defined as the concentration reached by the drug before the next dose administered. Data for this outcome measure was planned to be collected and analyzed separately for each dose of Teriflunomide. PK samples for teriflunomide 3.5 mg were collected during the first 8 weeks but all participants were switched to teriflunomide 7 mg after Week 8. Hence, plasma concentration of teriflunomide 7 mg and 14 mg were reported.
Time Frame: Predose on Week 36
Population: Analysis was performed on PK population which included all randomized participants exposed to DB study medication and had at least 1 PK sample taken. Here, 'overall number of participants analyzed' = participants evaluable for this outcome measure and "0'' signifies that none of the participant was evaluable for Teriflunomide 3.5 mg arm.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter
Groups:
- Teriflunomide 3.5 mg: Participants with BW up to 40 kg received 1 teriflunomide tablet, 3.5 mg orally once daily for 8 weeks. After 8 weeks, based on individual predicted PK parameters, teriflunomide was administered in following manner up to 96 weeks: if predicted PK parameters <= 95th percentile of adult range then participants received 1 tablet of 7 mg teriflunomide daily (for BW up to 40 kg) or 1 tablet of 14 mg teriflunomide daily (for BW >40 kg); or if predicted PK parameters >95th percentile of adult range then participants received 1 tablet of 3.5 mg teriflunomide daily (for BW <= 40 kg) or 1 tablet of 7 mg teriflunomide daily (for BW >40 kg).
- Teriflunomide 7 mg: Participants with BW >40 kg received 1 teriflunomide tablet, 7 mg orally once daily for 8 weeks. After 8 weeks, based on individual predicted PK parameters, teriflunomide was administered in following manner up to 96 weeks: if predicted PK parameters <= 95th percentile of adult range after 7 mg once daily then participants received 1 tablet of 7 mg teriflunomide daily (for BW up to 40 kg) or 1 tablet of 14 mg teriflunomide daily (for BW >40 kg); or if predicted PK parameters >95th percentile of adult range then participants received 1 tablet of 3.5 mg teriflunomide daily (for BW up to 40 kg) or 1 tablet of 7 mg teriflunomide daily (for BW >40 kg).
- Teriflunomide 14 mg: After 8 weeks, based on individual predicted PK parameters, teriflunomide was administered in following manner up to 96 weeks: if predicted PK parameters <= 95th percentile of adult range after 7 mg once daily then participants received 1 tablet of 7 mg teriflunomide daily (for BW up to 40 kg) or 1 tablet of 14 mg teriflunomide daily (for BW >40 kg); or if predicted PK parameters >95th percentile of adult range then participants received 1 tablet of 3.5 mg teriflunomide daily (for BW up to 40 kg) or 1 tablet of 7 mg teriflunomide daily (for BW >40 kg).
Arm/Group | Teriflunomide 3.5 mg | Teriflunomide 7 mg | Teriflunomide 14 mg
Number analyzed (Participants) | 0 | 10 | 66
micrograms per milliliter |  | 53.1 (25.3) | 67.8 (41.7)

21. Secondary Outcome: OL: Time to First Confirmed Clinical Relapse
Description: Time to first clinical relapse was defined as duration (in weeks) after enrollment in OL period and first confirmed clinical relapse. Clinical relapses were defined as new or recurrent neurological symptoms not associated with fever or infection, lasted at least 24 hours and accompanied by new objective neurological findings upon neurological examination and documented by standardized, quantified FSSs which included 8 items and items were rated on different scales: brain stem, cerebellar & cerebral functions rated on scale of 0 to 5; visual, pyramidal, sensory and bowel/bladder rated on scale of 0 to 6 and ambulation on scale of 0 to 12 where higher score in each scale indicated worsened neurological function. Confirmed clinical relapse were reviewed and confirmed by independent RAP. Participant without confirmed clinical relapse, was considered as clinical relapse free until end of Week 192.
Time Frame: Baseline up to Week 192
Population: Analysis was performed on efficacy population.
Measure: Median (Full Range); unit: weeks
Arm/Group | Placebo/Teriflunomide | Teriflunomide/ Teriflunomide
Number analyzed (Participants) | 52 | 100
weeks | 95.86 [0.6 to 176.0] | 96.00 [1.0 to 183.4]
Statistical Analysis 1: Comparison: Placebo/Teriflunomide vs Teriflunomide/ Teriflunomide; Test type: Other; Hazard Ratio (HR) = 0.693, 95% CI 2-sided [0.37 to 1.296] — Hazard ratio estimated using a Cox proportional-hazards model using treatment group, region, pubertal status, age, and number of relapses in the year prior to randomisation as covariates and with robust variance estimation

22. Secondary Outcome: OL: Pharmacokinetics: Steady-state Trough Concentration (Ctrough) of Teriflunomide
Description: Ctrough was defined as the concentration reached by the drug before the next dose is administered. Data for this outcome measure was planned to be collected and analyzed separately for each dose of teriflunomide. PK samples for teriflunomide 3.5 mg were collected during the first 8 weeks but all participants were switched to teriflunomide 7 mg after Week 8. Hence, plasma concentration of teriflunomide 7 mg and 14 mg were reported.
Time Frame: Pre-dose at Week 36
Population: Analysis was performed on PK population which included all randomized participants exposed to study medication, regardless of the amount of treatment administered who had at least one PK sample taken in OL period. Here, 'overall number of participants analyzed' = participants evaluable for this outcome measure and "0'' signifies that none of the participant was evaluable for Placebo/Teriflunomide 3.5 mg and Teriflunomide/Teriflunomide 3.5 mg arms.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter
Groups:
- Placebo / Teriflunomide 3.5 mg: Participants previously treated with placebo in DB period received 1 teriflunomide tablet 3.5 mg orally once daily for first 8 weeks of OL period. After 8 weeks, based on individual predicted PK parameters, teriflunomide was administered in following manner up to Week 192: if predicted PK parameters <= 95th percentile of adult range then participants received 1 tablet of 7 mg teriflunomide daily (for BW up to 40 kg) or 1 tablet of 14 mg teriflunomide daily (for BW >40 kg); or if predicted PK parameters >95th percentile of adult range then participants received 1 tablet of 3.5 mg teriflunomide daily (for BW up to 40 kg) or 1 tablet of 7 mg teriflunomide daily (for BW >40 kg).
- Placebo / Teriflunomide 7 mg: Participants previously treated with placebo during the DB period received teriflunomide 7 mg for 96 weeks in the OL period (i.e., up to Week 192).
- Placebo / Teriflunomide 14 mg: Participants previously treated with placebo during the DB period received teriflunomide 14 mg for 96 weeks in OL period (i.e., up to Week 192).
- Teriflunomide / Teriflunomide 3.5 mg: Participants previously treated with teriflunomide during the DB period received 1 teriflunomide tablet 3.5 mg orally once daily for first 8 weeks of OL period. After 8 weeks, based on individual predicted PK parameters, teriflunomide was administered in following manner up to Week 192: if predicted PK parameters <= 95th percentile of adult range then participants received 1 tablet of 7 mg teriflunomide daily (for BW up to 40 kg) or 1 tablet of 14 mg teriflunomide daily (for BW >40 kg); or if predicted PK parameters >95th percentile of adult range then participants received 1 tablet of 3.5 mg teriflunomide daily (for BW up to 40 kg) or 1 tablet of 7 mg teriflunomide daily (for BW >40 kg).
- Teriflunomide / Teriflunomide 7 mg: Participants previously treated with teriflunomide 7 mg during DB period continued receiving teriflunomide 7mg in the OL period for additional 96 weeks (i.e., up to Week 192).
- Teriflunomide / Teriflunomide 14 mg: Participants previously treated with teriflunomide 14 mg during DB period continued receiving teriflunomide 14mg in the OL period for additional 96 weeks (i.e., up to Week 192).
Arm/Group | Placebo / Teriflunomide 3.5 mg | Placebo / Teriflunomide 7 mg | Placebo / Teriflunomide 14 mg | Teriflunomide / Teriflunomide 3.5 mg | Teriflunomide / Teriflunomide 7 mg | Teriflunomide / Teriflunomide 14 mg
Number analyzed (Participants) | 0 | 12 | 31 | 0 | 2 | 79
micrograms per milliliter |  | 45.8 (35.3) | 50.4 (23.8) |  | 33.7 (10.7) | 63.6 (35.5)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs), treatment-emergent serious AEs and deaths were collected from first dose of study drug (Day 1) up to 96 weeks (for DB period arms), first dose of study drug in OL period (Week 97) up to Week 192 (for OL period arms) and first dose of study drug in extension period (Week 193) up to Week 492 (for extension period arm).
Description: Safety population included all randomized participants exposed to study medication, regardless of the amount of treatment administered.
Groups:
- Double-Blind Treatment Period: Placebo: Participants received placebo matching to teriflunomide tablet orally QD for 96 weeks.
- Double-Blind Treatment Period: Teriflunomide: Participants received 1 teriflunomide tablet, 3.5 mg (in case of BW up to 40 kg) or 7 mg (in case of BW >40 kg) orally QD for 8 weeks. After 8 weeks, based on participants predicted PK parameters, teriflunomide was administered in following manner up to 96 weeks: if predicted PK parameters <=95th percentile of adult range after 7 mg QD: 1 tablet of 7 mg daily (for BW up to 40 kg) or 1 tablet of14 mg daily (for BW>40 kg); or if predicted PK parameters >95th percentile of adult range:1 tablet of 3.5 mg daily (for BW up to 40 kg) or 1 tablet of 7 mg daily (for BW>40 kg). The adult range (5th-95th percentile) of predicted steady state PK parameters for 7 mg dose was defined as Cmax ranging from 8.03 to 49.10 mcg/mL and AUC0-24 ranging from 184 to 1160 mcg*h/mL.
- Open-Label Treatment Period: Placebo/Teriflunomide: Participants previously treated with placebo during the DB period received 1 teriflunomide tablet 3.5 mg (BW<=40 kg) or 7 mg teriflunomide (BW >40 kg) for first 8 weeks. After 8 weeks if predicted PK parameter was <= 95th percentile of adult range then participants received 7 mg teriflunomide (BW<=40 kg) and 14 mg teriflunomide (BW>40 kg) in the OL period for 96 weeks (i.e., up to Week 192). The adult range (5th-95th percentile) of predicted steady state PK parameters for 7 mg dose was defined as Cmax ranging from 8.03 to 49.10 mcg/mL and AUC0-24 ranging from 184 to 1160 mcg*h/mL.
- Open-Label Treatment Period: Teriflunomide/Teriflunomide: Participants previously treated with teriflunomide during DB period continued receiving teriflunomide in the OL period for additional 96 weeks (i.e., up to Week 192).
- Extension Period/Teriflunomide: Participants who were not adults when they completed the 192-week OL period were offered an optional additional extension period to receive 1 teriflunomide tablet 14 mg daily (or every other day if BW <40 kg) until they became adults or until they were able to switch to the commercial product, whichever came first.
Arm/Group | Double-Blind Treatment Period: Placebo | Double-Blind Treatment Period: Teriflunomide | Open-Label Treatment Period: Placebo/Teriflunomide | Open-Label Treatment Period: Teriflunomide/Teriflunomide | Extension Period/Teriflunomide
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/109 | 0/52 | 0/100 | 0/27
Serious Adverse Events (participants affected / at risk) | 6/57 | 12/109 | 15/52 | 14/100 | 8/27
Other Adverse Events (participants affected / at risk) | 42/57 | 89/109 | 40/52 | 72/100 | 18/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-Blind Treatment Period: Placebo (N=57) | Double-Blind Treatment Period: Teriflunomide (N=109) | Open-Label Treatment Period: Placebo/Teriflunomide (N=52) | Open-Label Treatment Period: Teriflunomide/Teriflunomide (N=100) | Extension Period/Teriflunomide (N=27)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Familial Mediterranean Fever (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sudden Hearing Loss (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anal Fissure (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal Fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Food Poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatic Disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis Acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gait Disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic Function Abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Complicated Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronavirus Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Encephalitis Viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary Tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Salpingo-Oophoritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Intentional Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint Dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral Nerve Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Blood Creatine Phosphokinase Increased (Investigations) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Transaminases Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Multiple Sclerosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Multiple Sclerosis Pseudo Relapse (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Multiple Sclerosis Relapse (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Partial Seizures (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 1 (1)
Transient Ischaemic Attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adjustment Disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Affective Disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression Suicidal (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Somatic Symptom Disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suicide Attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Renal Failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Drug Eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-Blind Treatment Period: Placebo (N=57) | Double-Blind Treatment Period: Teriflunomide (N=109) | Open-Label Treatment Period: Placebo/Teriflunomide (N=52) | Open-Label Treatment Period: Teriflunomide/Teriflunomide (N=100) | Extension Period/Teriflunomide (N=27)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 3 (3) | 0 (0) | 6 (6) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 3 (5) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 1 (1)
Sinus Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear Pain (Ear and labyrinth disorders) | 2 (2) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Autoimmune Thyroiditis (Endocrine disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye Pain (Eye disorders) | 4 (8) | 4 (4) | 0 (0) | 3 (3) | 0 (0)
Vision Blurred (Eye disorders) | 2 (3) | 2 (3) | 0 (0) | 3 (3) | 0 (0)
Visual Impairment (Eye disorders) | 2 (3) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 11 (13) | 2 (2) | 8 (11) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 2 (2) | 6 (9) | 0 (0) | 3 (4) | 0 (0)
Aphthous Ulcer (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 3 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 8 (9) | 6 (8) | 7 (9) | 1 (1)
Gastrointestinal Disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mouth Ulceration (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (4) | 2 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (5) | 10 (12) | 3 (3) | 4 (4) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (3) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (5) | 6 (7) | 2 (2) | 2 (2) | 0 (0)
Asthenia (General disorders) | 0 (0) | 2 (2) | 2 (3) | 1 (1) | 0 (0)
Fatigue (General disorders) | 3 (5) | 4 (6) | 4 (7) | 4 (4) | 0 (0)
Influenza Like Illness (General disorders) | 1 (1) | 3 (3) | 0 (0) | 2 (2) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 4 (4) | 0 (0) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 5 (8) | 0 (0) | 3 (3) | 2 (2)
Acute Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 5 (5) | 2 (2) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Cystitis (Infections and infestations) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (3) | 3 (3) | 2 (2) | 5 (6) | 1 (1)
Influenza (Infections and infestations) | 4 (4) | 10 (16) | 5 (6) | 5 (6) | 2 (3)
Nasopharyngitis (Infections and infestations) | 5 (6) | 28 (50) | 8 (13) | 20 (37) | 4 (4)
Paronychia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 7 (8) | 1 (2) | 4 (8) | 1 (1)
Pulpitis Dental (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory Tract Infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 5 (5) | 1 (1)
Respiratory Tract Infection Viral (Infections and infestations) | 0 (0) | 4 (7) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 2 (3) | 4 (8) | 2 (4) | 6 (7) | 1 (1)
Root Canal Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2) | 4 (4) | 2 (3) | 2 (2) | 0 (0)
Tinea Versicolour (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 2 (2) | 4 (4) | 2 (4) | 4 (5) | 0 (0)
Tracheitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Tracheobronchitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 6 (23) | 24 (66) | 7 (32) | 22 (59) | 6 (12)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 3 (3) | 2 (2) | 5 (5) | 0 (0)
Accidental Overdose (Injury, poisoning and procedural complications) | 4 (7) | 5 (5) | 2 (2) | 10 (12) | 3 (3)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 4 (4) | 1 (1) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 4 (5) | 6 (8) | 2 (3) | 1 (1) | 0 (0)
Hip Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ligament Sprain (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 1 (3) | 2 (2) | 0 (0)
Thermal Burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 1 (1) | 2 (3) | 6 (6) | 3 (3) | 2 (2)
Aspartate Aminotransferase Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Blood Albumin Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood Bilirubin Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood Creatine Phosphokinase Increased (Investigations) | 0 (0) | 4 (6) | 1 (1) | 0 (0) | 2 (2)
Blood Uric Acid Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram St-T Segment Abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gamma-Glutamyltransferase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Glomerular Filtration Rate Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematocrit Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haemoglobin Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Monocyte Count Decreased (Investigations) | 0 (0) | 1 (2) | 1 (1) | 3 (4) | 0 (0)
Monocyte Percentage Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil Count Decreased (Investigations) | 0 (0) | 3 (5) | 1 (4) | 2 (6) | 3 (5)
Neutrophil Percentage Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil/Lymphocyte Ratio Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Protein Urine Present (Investigations) | 1 (1) | 4 (5) | 2 (2) | 1 (1) | 0 (0)
Weight Decreased (Investigations) | 3 (3) | 6 (7) | 2 (2) | 3 (5) | 0 (0)
Weight Increased (Investigations) | 0 (0) | 3 (4) | 0 (0) | 2 (3) | 0 (0)
White Blood Cell Count Decreased (Investigations) | 1 (1) | 5 (8) | 2 (5) | 5 (9) | 3 (7)
White Blood Cells Urine Positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 0 (0) | 3 (3) | 1 (1)
Iron Deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitamin D Deficiency (Metabolism and nutrition disorders) | 2 (2) | 3 (4) | 1 (1) | 4 (4) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (7) | 5 (5) | 2 (2) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 5 (6) | 2 (3) | 3 (5) | 0 (0)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 0 (0) | 3 (4) | 0 (0)
Disturbance In Attention (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 4 (5) | 9 (9) | 6 (12) | 2 (3) | 0 (0)
Headache (Nervous system disorders) | 13 (18) | 18 (30) | 7 (22) | 14 (28) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 3 (5) | 6 (7) | 3 (4) | 3 (4) | 1 (1)
Paraesthesia (Nervous system disorders) | 2 (3) | 11 (19) | 1 (1) | 4 (7) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 2 (3) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 3 (3) | 4 (6) | 1 (1) | 2 (3) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 2 (2) | 4 (4) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (3) | 1 (1) | 1 (3) | 1 (1) | 0 (0)
Mixed Anxiety And Depressive Disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Micturition Urgency (Renal and urinary disorders) | 1 (1) | 2 (2) | 5 (6) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 3 (3) | 1 (1) | 1 (4) | 2 (5) | 1 (1)
Menstrual Disorder (Reproductive system and breast disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (6) | 2 (2) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (4) | 0 (0) | 1 (3) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 7 (8) | 2 (2) | 7 (9) | 1 (1)
Respiratory Disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 4 (4) | 5 (5) | 0 (0) | 4 (5) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 7 (7) | 24 (26) | 9 (10) | 10 (10) | 1 (1)
Dry Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (4) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4) | 2 (2) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (5) | 1 (1)
Orthostatic Hypotension (Vascular disorders) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2020-12-10): https://cdn.clinicaltrials.gov/large-docs/08/NCT02201108/Prot_002.pdf
  • Statistical Analysis Plan (2021-06-28): https://cdn.clinicaltrials.gov/large-docs/08/NCT02201108/SAP_003.pdf